CLINICAL TRIAL: NCT06322563
Title: An Open, Single-arm, Phase II Clinical Study Evaluating the Safety and Initial Efficacy of LTC004 in Combination With Regorafenib in the Treatment of Metastatic Colorectal Cancer
Brief Title: Combination of LTC004 and Regorafenib to Treat Patients With Advanced/Metastatic CRC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LTC004-202
Record Dates: First submitted 2024-02-26; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-02

CONDITIONS: Advanced/Metastatic Colorectal Cancer
Keywords: mCRC
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety introduction trial：LTC004+regorafenib (Experimental): LTC004 in combination with regorafenib safety introduction trial and completing a 28-day safety assessment
  Interventions: Drug: LTC004+regorafenib
- Formal trial phase：LTC004+regorafenib (Experimental): After Safety introduction trial, safety will be confirmed before entering the formal trial phase.Further evaluation of the safety and efficacy of LTC004 in combination with regorafenib in the treatment of mCRC
  Interventions: Drug: LTC004+regorafenib

INTERVENTIONS:
Drug: LTC004+regorafenib — LTC004,90μg/kg,IV,Day 1,Q3W; Regorafenib:Orally once daily for the first 21 days of each cycle, with 28 days as 1 cycle. Cycle 1 was dose-escalation with a starting dose of 80 mg/d, increasing by 40 mg per week until 160 mg/d, i.e., 80 mg/d in week 1 (D1~D7), 120 mg/d in week 2 (D8~D14), and 160 mg/d in week 3 (D15~D21);

SUMMARY:
This is a phase II clinical study to evaluate the safety, tolerability and preliminary antitumor activity of LTC004 in combination with regorafenib in patients with mCRC. A safety introductory trial was conducted to receive LTC004 in combination with regorafenib before starting the formal trial. After completing a 28-day safety assessment, safety will be confirmed before entering the formal trial phase. Further evaluation of the safety and efficacy of LTC004 in combination with regorafenib in the treatment of mCRC

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years.
2. Non-radical resectable metastatic colorectal cancer confirmed by histology or cytology.
3. Those who have progressed on, or are intolerant to, at least one prior first- and second-line systemic antitumor therapy for metastatic colorectal cancer. Patients must have received fluorouracil, oxaliplatin, and irinotecan-based chemotherapy, and patients with mCRC who have previously received or are not candidates for anti-VEGF therapy, anti-epidermal growth factor receptor therapy (RAS wild-type).
4. Pre-existing MMR, MSS, HER2, PD-L1, RAS, and BRAF status with corresponding supporting documentation.
5. At least one measurable tumor lesion based on RECIST V1.1 criteria.
6. ECOG PS ≤1.
7. Expected survival ≥12 weeks.
8. able to Swallow whole pills.
9. Adequate organ function.
10. Patients, both females and males, of reproductive potential must agree to use adequate contraception during and for 6 months after the last infusion of LTC004.
11. Understands and provides written informed consent and willing to follow the requirements specified in protocol.

Exclusion Criteria:

1. History of severe hypersensitivity reactions to other mAbs.
2. Untreated, unstable or uncontrolled central nervous system (CNS) metastases.
3. Tumor invasion of vital arteries resulting in high risk of bleeding, significant risk of perforation or already formed fistulae.
4. Patients with uncontrolled pleural effusion, pericardial effusion or abdominal effusion as judged by the investigator at screening.
5. Patients with untreated or clinically symptomatic spinal cord compression that has not been controlled.
6. Previous antitumor regimens include immunotherapies such as PD-1/L1 inhibitors, LAG3, TIGIT, IL-2, IL-15, CD3-like immunoagonists, and other cellular therapies, as well as other TKI agents (e.g., furaquintinib, regorafenib, etc.).
7. ≥2 malignant tumors within 5 years prior to first dose of drug.
8. Patients who have received any chemotherapy or anti-tumor monoclonal antibody drugs within 4 weeks prior to the first dose of study drug (excluding mitomycin and nitrosoureas within 6 weeks prior to the first dose of study drug; small molecule targeted drugs within 2 weeks prior to the first dose of study drug; Chinese medicine therapy (Chinese medicine therapy with clear anti-tumor indications in the package insert within 4 weeks prior to the first dose of study drug.
9. Moderate to severe dyspnea at rest due to advanced cancer or its complications, severe primary lung disease, current need for continuous oxygen therapy, or clinically active interstitial lung disease (ILD) or pneumonia; Grade ≥3 interstitial pneumonia during prior antineoplastic therapy.
10. Presence of severe infections including, but not limited to, bacteremia and severe pneumonia requiring hospitalization within 4 weeks prior to the first dose; active infections with CTCAE ≥ grade 2 requiring treatment with systemic antibiotics within 2 weeks prior to the first dose.
11. History of serious cardiovascular disease.
12. Previous total gastrectomy, chronic diarrhea, active inflammatory gastrointestinal disease, or any other condition causing malabsorption syndrome.
13. Active bleeding disorder, including gastrointestinal bleeding, as evidenced by vomiting of blood, profuse hemoptysis, or black stools, in the 6 months prior to enrollment.
14. Active hepatitis B (hepatitis B virus DNA measurement ≥1000 copies/mL or 200 IU/mL); hepatitis C infection (hepatitis C antibody positive and HCVRNA above the lower limit of detection in research centers); syphilis infection, active tuberculosis.
15. Active, or previous autoimmune disease with potential for recurrence at the time of screening.
16. Immunodeficiency diseases or history of such diseases, including a positive serologic test for human immunodeficiency virus (HIV).
17. Arterial/venous thrombotic events within 6 months prior to first dose.
18. Those who received radical radiation therapy within 4 weeks prior to the first dose and those who received palliative radiation within 14 days prior to the first dose.
19. Use of live or attenuated vaccines within 4 weeks prior to the first dose, or anticipated need for live or attenuated vaccines during the study period.
20. Major surgery (other than surgery for diagnostic purposes) within 4 weeks prior to the first dose, anticipation of major surgery (other than surgery for diagnostic purposes) during the study period, or diagnostic or low-invasive surgery within 7 days prior to the first dose (excluded for puncture biopsy).
21. Adverse effects of prior antineoplastic therapy have not returned to a CTCAE version 5.0 grade rating of ≤ grade 1 (with the exception of alopecia and grade 2 neurotoxicity due to chemotherapeutic agents, and grade 2 hypothyroidism due to antineoplastic therapy).
22. Patients with prior allogeneic bone marrow/hematopoietic stem cell transplantation or solid organ transplantation.
23. Pregnant, lactating women.
24. Subjects who, in the judgment of the investigator, have a history of other serious systemic disease or are unfit to participate in this trial for any other reason (the presence of psychiatric disorders in the patient that may affect compliance with the trial, alcohol, drug or substance abuse, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events-Safety and Tolerability | up to 12 months
  TEAE and changes in safety indicators (12-ECG,Laboratory inspection items,Cardiopulmonary function and so on)before and after administration
SAE-Safety and Tolerability | up to 12 months
  SAE and changes in safety indicators (12-ECG,Laboratory inspection items,Cardiopulmonary function and so on)before and after administration

SECONDARY OUTCOMES:
ORR | up to 12 months
  Antitumor efficacy of LTC004+Regorafenib
DCR | up to 12 months
  Antitumor efficacy of LTC004+Regorafenib
PFS | up to 12 months
  Antitumor efficacy of LTC004+Regorafenib
OS | up to 12 months
  Antitumor efficacy of LTC004+Regorafenib

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No